CLINICAL TRIAL: NCT05221138
Title: A Phase I Clinical Trial to Evaluate the Food Effect on Pharmacokinetic Profiles of VV116 Administered Orally to Chinese Healthy Volunteers
Brief Title: Food Effect on Pharmacokinetic Profiles of VV116 Administered Orally to Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VV116-03
Record Dates: First submitted 2021-12-29; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Healthy Subjects
Keywords: VV116; three-period crossover; food effect
MeSH Terms: interventions — GS-621763

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VV116 after High-fat meal intake (Experimental): a single oral after High-fat meal intake
  Interventions: Drug: VV116
- VV116 after Fasting+Standard diet (Experimental): a single oral after Fasting
  Interventions: Drug: VV116
- VV116 after Standard meal intake (Experimental): a single oral after Standard meal intake
  Interventions: Drug: VV116

INTERVENTIONS:
Drug: VV116 — VV116 oral tablets, 400mg

SUMMARY:
This study is a single-center, randomized, open-label, three-period crossover design, the objective is to evaluate the pharmacokinetics and safety of VV116 tablets, which are orally administered to Chinese healthy volunteers after fasting, standard diet or high-fat diet.

DETAILED DESCRIPTION:
12 healthy subjects will be enrolled once all eligibility criteria are met after screening within 14 days prior to investigation product administration. Informed consent should be obtained before any protocol defined procedures can be started.

Investigational product administration plan given below: 12 healthy subjects will be randomized to 3 groups, i.e., Group A, Group B, Group C, with 4 subjects in each group. For group A, investigation product will be given after fasting for Period 1, after standard diet for Period 2, and after high-fat diet for Period 3; For group B, investigation product will be given after high-fat diet for Period 1, after fasting for Period 2, and after standard diet for Period 3; For group C, investigation product will be given after standard diet for Period 1, after high-fat diet for Period 2, and after fasting for Period 3. Wash-out period is 3 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects between the ages of 18 and 45 years;
2. Body weight no less than 50 kg for male, no less than 45 kg for female; Body Mass Index of 19 to 26kg/m2;
3. Physical examination, vital signs examination, laboratory examination, ECG, B-ultrasound and fundus examination results were normal or abnormal without clinical significant;
4. Subjects who are willing to take proper contraceptive during the study and within 3 months after the study completed;
5. Subjects who are able to understand and follow study plans and instructions; Subjects who have voluntarily decided to participate in this study, and signed the informed consent form;

Exclusion Criteria:

1. Subjects with hypersensitivity to VV116 or any of the excipients;
2. Subjects with allergic diseases or allergic constitution;
3. Subjects with central nervous system,cardiovascular system,gastrointestinal, respiratory system,urinary,Hematologic System,metabolic disorders that require medical intervention or other diseases (such as psychiatric history) that are not suitable for clinical trials;
4. Blood donation or blood loss ≥ 400 mL within 3 months prior to inclusion, or have a history of blood product use history;
5. Participated in a clinical study involving another investigational drug within 3 month before the screening visit;
6. Taken any prescription drugs, non-prescription drugs, Chinese herbal medicine or health care products within 2 weeks prior to screening;
7. Drug or alcohol addicts within 1 year prior to screening, who drink at least twice a day or more than 14 units per week, or who are addicted to alcohol (1 unit ≈200 mL beer with 5% alcohol content, 25 mL spirits with 40% alcohol content or 85 mL wine with 12% alcohol content) ;
8. Those who smoke more than 10 cigarettes per day and do not agree to avoid using any tobacco products during the trial period;
9. Those who cannot quit smoking or drinking during the trial;
10. Those who are positive for hepatitis B surface antigen (HBsAg), HCV antibody, syphilis antibody and HIV antibody;
11. Abnormal and clinically significant chest radiographs (anteroposterior);
12. B ultrasound examination showed moderate to severe fatty liver;
13. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeded the upper normal limit (ULN) at screening time or baseline;
14. Glomerular filtration rate (eGFR) < 90 mL/min/1.73m2 at screening time or baseline;
15. Abnormal ecg at screening or baseline, single QTcF (corrected for heart rate) > 450 ms in men, > 470 ms in women, and/or other clinically significant abnormalities;
16. Pregnant or lactating women or male subjects whose spouse has a child care plan within 3 months;
17. The investigator believes that there are other factors that are not suitable for participating in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Evaluate high-fat diet and standard diet's effect on Cmax of VV116 tablets | From time zero up to 48 hours post-dose following oral administration of VV116
  maximum observed plasma concentration
Evaluate high-fat diet and standard diet's effect on AUC0-t of VV116 tablets | From time zero up to 48 hours post-dose following oral administration of VV116
  area under the plasma concentration time curve from time zero to the last measurable concentration
Evaluate high-fat diet and standard diet's effect on AUC0-∞ of VV116 tablets | From time zero up to 48 hours post-dose following oral administration of VV116
  area under the plasma concentration-time curve from time zero to infinity
Evaluate high-fat diet and standard diet's effect on Tmax of VV116 tablets | From time zero up to 48 hours post-dose following oral administration of VV116
  time at which Cmax occurs

SECONDARY OUTCOMES:
The incidence and severity of treatment emergent adverse event (TEAE) of clinical symptoms | 7 days after last treatment
  The incidence and severity of treatment emergent adverse event (TEAE), including Serious Adverse Event (SAE), as well as clinical symptoms, and any abnormalities of vital signs, physical examinations, , ophthalmology and, etc.
The incidence and severity of treatment emergent adverse event (TEAE) of vital signs | 7 days after last treatment
  The incidence and severity of treatment emergent adverse event (TEAE) of vital signs
The incidence and severity of treatment emergent adverse event (TEAE)of physical examinations | 7 days after last treatment
  The incidence and severity of treatment emergent adverse event (TEAE)of physical examinations
The incidence and severity of treatment emergent adverse event (TEAE) of laboratory tests | 7 days after last treatment
  The incidence and severity of treatment emergent adverse event (TEAE) of laboratory tests
The incidence and severity of treatment emergent adverse event (TEAE) of physical examinations | 7 days after last treatment
  The incidence and severity of treatment emergent adverse event (TEAE) of physical examinations
The incidence and severity of treatment emergent adverse event (TEAE) of electrocardiogram (ECG) | 7 days after last treatment
  The incidence and severity of treatment emergent adverse event (TEAE) of electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Gangyi Liu, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No